CLINICAL TRIAL: NCT04966156
Title: A Longitudinal Multidimensional Cancer Rehab Program for Patients Undergoing Allogenic Bone and Marrow Transplantation (CaRE-4-alloBMT)
Brief Title: Cancer Rehab Program for Allogenic Bone and Marrow Transplant Patients - CaRE-4-alloBMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 21-5076.0
Record Dates: First submitted 2021-04-26; First posted 2021-07-19 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Allogeneic Disease; Hematologic Cancer; Cancer Rehabilitation
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be informed when consented that they will be grouped into one of two (control or intervenion) study groups for the duration of the study. Following their baseline assessment, patients will be randomized (1:1 stratified by age and clinical frailty score at pre-transplant consultation).
Who Masked: Participant
Masking Description: biostatician will provide the randomized grouping for each of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care group (No Intervention): No change to patient's usual care at Princess Margaret Cancer Centre.
- CaRE-4-allBMT plus usual care (Experimental): a longitudinal 6-month rehabilitation program that uses a person- centred strategy and a multidimensional approach targeting physical activity, nutrition, psychosocial distress and promoting self-management skills.
  Interventions: Behavioral: CaRE-4-alloBMT plus usual care group

INTERVENTIONS:
Behavioral: CaRE-4-alloBMT plus usual care group — CaRE-4-alloBMT uses emerging eHealth technologies to reduce barriers to accessing and providing cancer rehabilitation which includes: 1) Individualized progressive exercise prescriptions that allows customizable exercise prescriptions, tracking of exercise completion, and video tutorials; 2) Individualized nutrition plans and stepped stratified care such as education, counselling, intervention based on nutritional status and delivered by registered dietitians; 3) On-line e-modules provide interactive education to promote self-management skills for stress management, nutrition, managing common symptoms, etc.; 4) Remote monitoring using FitbitTM devices to monitor patients physical activity, caloric intake, and sleep for duration of the program. CRS and alloBMT clinicians will have access to real-time Fitbit data through our clinical dashboard; 5) Remote clinical support: check-ins and health coaching sessions with a member of the CRS team (phone or MS Teams video).
  Arms: CaRE-4-allBMT plus usual care

SUMMARY:
Currently, transplantation centers across North America generally do not offer longitudinal rehabilitation programs and research is urgently needed to test the acceptability and effectiveness of these programs using innovative delivery strategies that have the potential for future scalability and to understand the associated costs. Through a strong collaboration between the PM Cancer Rehabilitation and Survivorship (CRS) and alloBMT teams, the principal investigators developed an innovative multicomponent rehabilitation intervention for patients undergoing alloBMT (CaRE-4-alloBMT).

CaRE-4-alloBMT uses a person- centred strategy and a multidimensional approach targeting physical activity, nutrition, psychosocial distress and promoting self-management skills. Innovative components of CaRE-4-alloBMT include:1) Individualized progressive exercise prescriptions developed and monitored by CRS registered kinesiologists and supported with a web/mobile application (Physitrack) that allows customizable exercise prescriptions, tracking of exercise completion, and video tutorials; 2) Individualized nutrition plans and stepped stratified care (education, counselling, intervention) based on nutritional status and delivered by registered dietitians (alloBMT and CRS). 3) On-line e-modules (developed in collaboration with PM Oncology Education) provide interactive education to promote self-management skills on crucial topics; 4) Remote monitoring using FitbitTM devices to monitor patients physical activity, caloric intake, and sleep for duration of the program; 5) Remote clinical support: Pre/Post discharge, patients will have scheduled (PHS) remote check-ins and health coaching sessions with a member of the CRS team (phone or MS Teams video).

Objectives: i) To test the feasibility and safety of CaRE-4-alloBMT plus standard best practice cancer care compared to standard best practice cancer care alone; ii) To assess the preliminary efficacy of CaRE-4-alloBMT on physical function, disability, nutritional status, distress, QoL, healthcare utilization, and survival and estimate program return on investment.

DETAILED DESCRIPTION:
1.0 BACKGROUND: Allogeneic blood and marrow transplantation (alloBMT) is a curative treatment for many hematologic cancers and its use has increased rapidly over the past decade. While effective, alloBMT is associated with numerous treatment-related physical and psychosocial side effects, reduced physical functioning, and worsening nutritional status which are associated with increased risk of complications (i.e. infections, drug toxicity, weight loss, graft failure & graft-versus-host disease), significant early and late treatment related mortality, and can profoundly affect quality of life (QoL).

As a result, there have been calls for increased attention to the management of adverse effects associated with alloBMT with the goal to minimize dysfunction, maximize well-being and QoL, and reduce treatment-related mortality.

Cancer rehabilitation is now considered an essential component of cancer care and focuses on prevention and treatment of the adverse effects of cancer and treatment and to optimize functional status and QoL. Embedding multidimensional longitudinal (pre to post transplant) rehabilitation programs that focus on exercise, nutrition and teaching self-management skills as a standard part of treatment for individuals undergoing alloBMT has potential to mediate the significant adverse effects, improve survival, and reduce burden on the healthcare system. While patients typically receive some in-patient rehabilitation, this is a small part of the alloBMT pathway and services are quite limited. Currently, transplantation centers across North America generally do not offer longitudinal rehabilitation programs and research is urgently needed to test the acceptability and effectiveness of these programs using innovative delivery strategies that have the potential for future scalability and to understand the associated costs. In response, through a strong collaboration between the PM Cancer Rehabilitation and Survivorship (CRS) and alloBMT teams, the principal investigators developed an innovative multicomponent rehabilitation intervention for patients undergoing alloBMT (CaRE-4-alloBMT).

2.0 PROGRAM DESCRIPTION (see Appendix 1): CaRE-4-alloBMT is a longitudinal 6-month rehabilitation program (peri to post transplant) adapted from an existing evidence-based and effective model developed by the CRS team (CaRE@ELLICSR and CaRE@Home). The program is informed by established behaviour change theory and harnesses current and emerging eHealth technologies to reduce barriers to accessing and providing cancer rehabilitation. CaRE-4-alloBMT uses a person- centred strategy and a multidimensional approach targeting physical activity, nutrition, psychosocial distress and promoting self-management skills. Innovative components of CaRE-4-alloBMT include:

1. Individualized progressive exercise prescriptions developed and monitored by CRS registered kinesiologists and supported with a web/mobile application (Physitrack) that allows customizable exercise prescriptions, tracking of exercise completion, and video tutorials. The initial personalized exercise program will be given to a participant following the initial assessment. A program will be created based on the specific needs and physical condition of each participant. The participant will receive the detailed exercise program via Physitrack (includes exercise description and videos of each exercise). Each exercise program will contain cardiovascular and strength training as well as stretching exercises. The exercise program will be revised and progressions will be added based on the individual's needs after the follow-up assessments or during the scheduled check-ins between assessments. Check-ins are scheduled as follows:

   * At 2 and 4 weeks after initial assessment
   * 8 weekly check-ins following discharge
   * At 10 and 12 weeks following discharge The participant can contact the Kinesiologist by e-mail at any point during the program.
2. Individualized nutrition plans and stepped stratified care (education, counselling, intervention) based on nutritional status and delivered by registered dietitians (alloBMT and CRS). As part of standard of care, all patients receive a nutrition assessment and their caloric intake goals are set. Those in the INT arm (CaRE-4-alloBMT plus usual care group) will receive additional nutritional education through the e-modules and monitoring of caloric intake through the Fitbit. They will also have access to meal preparation and recipes through ellicsrkitche.ca. Patients can track their nutritional intake on their Fitbit device and this data will be monitored weekly by the RKin. Patients who falls below 50% of their goals (based on intake assessment) will flagged to the RD for follow up.
3. On-line e-modules (developed in collaboration with PM Oncology Education) provide interactive education to promote self-management skills on crucial topics (i.e. stress management, nutrition, managing common symptoms). There will be 9 online e-modules:

   * Introduction: Getting started
   * Eat and Cook for Wellness
   * Exercise
   * Manage Your Emotions
   * Reduce Fatigue
   * Being Mindful
   * Boost Your Brain Health
   * Stay Connected
   * Planning for the Future Participants will be asked to complete all 9 modules. Each module should take between 20-30 minutes to complete. Participants can go through these modules at their own pace. Patients will receive a link for the online modules. Patients will be able to access the module by entering their e-mail address and creating their own unique password.
4. Remote monitoring using FitbitTM devices to monitor patients physical activity, caloric intake, and sleep for duration of the program. CRS and alloBMT clinicians will have access to real-time Fitbit data through the clinical dashboard (developed in collaboration with TECHNA). The Fitbit is also known to promote behaviours change and allows for self-monitoring and feedback. Participants will be asked to wear the Fitbit for the duration of the study. Participants will only need to add their meals to monitor their nutrition. No other action is required from the participants once the account has been created. This will replace the paper based food diary they must keep (standard of care). The account for the participant will be created by the RA or RKin and the participant will then be able to access the app via an email link. The RA or RKin can assist/provide support to the participant as needed to access the app. If the participant is unable to download or use the app a detailed print out of their exercise program will be provided.

   The following information will be required to create an account:
   * First name
   * Last name (participant study number will be entered in this field
   * Year of birth
   * Email address Both the participant and Kinesiology team will have access to this information but the account information is not visible to third parties. Physitrack provides links to the privacy policy and terms of use/agreement and is available for the participant to review as needed.
5. Remote clinical support: Pre/Post discharge, patients will have scheduled (PHS) remote check-ins and health coaching sessions with a member of the CRS team (phone or MS Teams video). These occur in week 2,4 (pre) and 1-8,10,12 (post-discharge).

Frequency of check-ins and what will be discussed: Check-ins are by telephone or MSteams video and scheduled as follows:

* At 2 and 4 weeks after initial assessment (pre-BMT admission)
* Weeks 1-8, 10 and 12 post-discharge (post-BMT dischange)

  - Check-ins discussion using motivational interviewing techniques and focus on
* Adherence to exercise program
* Changes to exercise program based on participant's needs
* Module completion
* Answering participants questions The program strongly aligns with the SUNDAE framework

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Must have received a hematologic cancer diagnosis
* Awaiting alloBMT
* Able to communicate in English
* Able to access online study material (Physitrack and education e-modules).

Exclusion Criteria:

* Not meeting the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-09-08 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Drop-out rates as a measure of feasibility | 6 months
  Number of patients who complete the study/ drop-out will be used to identify feasibility of the intervenion.
Patient preference as assessed during clinical support as a measure of feasibiity | 6 months
  Check-ins with health coach during assessments will be used to identify intervention acceptability/preference.
Measuring safety as assessed during one-on-one interviews with health coach - this wll be (analyzed as qualitative data) done over MS Teams and will be a conversational question and answer format. | 6 months
  Patients will be checking-in at specific timepoints with a health coach to discuss their preference/challenges with intervention.

SECONDARY OUTCOMES:
Disability assessment schedule | 6 months
  World Health Organization Disability Assessment Schedule 2.0. The scale is (0-4) for a total score from 0-48 and the larger the value the worse the outcome.
36 items short form health survey | 6 months
  self reported measure of overall health - total score: 0-100 and the higher the score, the better the health state (less disability)
Evaluating nutritional status based on caloric intake | 6 months
  using data from fitbit worn by patient to record their daily caloric intake.
Using the Body Mass Indext to measure nutritional status | 6 months
  Body Mass Index
Measure of nutritional status by using the Patient Generated Subjective Global Assessment | 6 months
  Patient-reported instrument for assessment of nutrition status in patients with cancer - Typical scores range from 0-35 with a higher score reflecting a greater risk of malnutrition and scores ≥9 indicating a critical need for nutrition intervention and symptom management.
General Anxiety Disorder assessment | 6 months
  Measure of General Anxiety and distress - total score: 0-21 and the cut-offs are: 0-4: minimal anxiety 5-9: mild anxiety 10-14: moderate anxiety 15-21: severe anxiety
Functional Assessment of Cancer Therapy for Bone Marrow Transplant | 6 months
  a measure of quality of life - total score of 0-196 with a higher scores for the scales and subscales indicate better quality of life.
Measure of the level of healthcare utilization by patient | 6 months
  clinic chart details for days in hospital, readmission
measure of overall survival | 6 months
  will be interpretted from the quantitative and qualitative date extracted
Euroqol 5D | 6 months
  Health related quality of life - The maximum score of 1 indicates the best health state, by contrast with the scores of individual questions, where higher scores indicate more severe or frequent problems.
6 minute walk test | 6 months
  measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface
grip strength tests | 6 months
  measures the muscular strength or the maximum force/tension generated by one's forearm muscles
Sit-to-stand test | 6 months
  measurement that assesses functional lower extremity strength in older adults

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M Jones, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tam S, Alibhai SMH, Hassanieh D, Kumar R, Mattsson J, Atenafu EG, Avery L, Bernstein LJ, Chang E, Langelier D, Lopez P, Jones JM. A phase 2 study of a longitudinal multidimensional rehabilitation program for allogeneic blood and marrow transplantation patients. Blood Adv. 2024 Sep 24;8(18):4778-4791. doi: 10.1182/bloodadvances.2024012968. PMID 38985303